CLINICAL TRIAL: NCT00669513
Title: Cardiovascular Effects of Partial Sleep Deprivation in Healthy Volunteers
Brief Title: Cardiovascular Effects of Partial Sleep Deprivation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PSP-CV
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Sleep Deprivation
Keywords: partial sleep deprivation; endothelial dysfunction; sympathetic activity; inflammation
MeSH Terms: conditions — Sleep Deprivation; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Partial sleep deprivation
  Interventions: Behavioral: Partial sleep deprivation

INTERVENTIONS:
Behavioral: Partial sleep deprivation — Partial sleep deprivation (less than 5 hours, but no less than 3 hours and 30 minutes)
  Arms: 2

SUMMARY:
Background: Sleep curtailment is common and is associated with increased mortality due to cardiovascular causes. However, the mechanisms are not completely understood.We hypothesized that partial sleep deprivation caused however significant changes in sympathetic activity and endothelial function in healthy volunteers.

Methods: Thirteen young healthy male volunteers will be monitored during 12 days by sleep diary and wrist actigraphy. The subjects will keep under their usual daily activities and randomized to 5 nights of prolonged sleep (control) or partial sleep deprivation, interposed by 2 nights of unrestricted sleep (wash out). At the end of each period, the subjects will be evaluate by: 1. electrocardiogram and beat-to-beat blood pressure with spectral analysis of heart rate and blood pressure in the supine position and after head up tilt test maneuver; 2. resting plasma norepinephrine; 3. venous endothelial function (dorsal hand vein technique).

DETAILED DESCRIPTION:
Volunteers Healthy young male volunteers from the urban area of Sao Paulo city will be recruited to the study. All subjects will be clinically evaluated, including measurements of weight and height. Exclusion criteria include age less than 21 and more than 45 years, body mass index (BMI) >25 kg/m2, smoking, use of chronic medications and any established medical condition including diabetes mellitus, hypertension, dyslipidemia, heart diseases and sleep disordered breathing. After obtaining written informed consent, all participants will be submitted to overnight polysomnography.

Polysomnography Overnight polysomnography will be performed to discarded sleep breathing using a digital system (17 channels, EMBLA Medicare - Flaga hf. Medical Devices). All polysomnograms will be performed and scored based on the guidelines for sleep studies. The apnea-hypopnoea index (AHI) was defined by the number of apneas and hypopnoeas per hour of sleep. Sleep disordered breathing was defined by an AHI above 5 events/hour, according to standard criteria.

Sleep Monitoring During the study period all subjects will be continuously monitored by a sleep diary and wrist actigraphy (Basic Mini Motionlogger Actigraph Ambulatory Monitoring, Inc., Ardsley , New York, USA ) worn on the non-dominant hand. The actigraph will set to sample movements in 1 min periods. Actigraph records will automatically process by use of the AW2 software version 2.3.01 program (Ambulatory Monitoring, Inc.) to extract information on sleep duration.

Blood Samples Venous blood will be collected from all participants between 8 and 10 AM for the measurement of glucose, total cholesterol, low-density lipoprotein, high-density lipoprotein, and red blood cell count. Plasma catecholamine (norepinephrine) will be measured by High-Performance Liquid Chromatography.

Hemodynamic and autonomic measurements Hemodynamic and autonomic evaluations will be performed in the morning between 8 and 10 AM. The intervals between adjacent QRS complexes resulting from sinus node depolarization will be determined (RR intervals). Heart rate will be calculated by expressing RR intervals as beats per minute. Non-invasive beat-to-beat blood pressure (Finometer, Finapres Medical System BV, Holland) and electrocardiogram (ECG) will be continuously recorded by the software AT/MCA-CODAS (DATAC Instruments Inc., Akron, Ohio, EUA). The sampling rate was 1000 Hz per channel.

Autonomic measurements will be derived from spectral analysis of HR and systolic blood pressure (SBP). For frequency domain analysis, power spectral density will be obtained by the Fast Fourier Transformation using the Welch's method over 16,384 points with a Hanning window (512) and 50% overlapping. Spectral power for low- (LF 0.04-0.15 Hz), and high- (HF 0.15-0.4 Hz) frequency bands will be calculated by means of power spectrum density integration within each frequency bandwidth, using a customized routine (MATLAB 6.0, Mathworks). LF/HF ratio will be also calculated to evaluate the sympathovagal balance. In addition, we will also evaluated the power spectral analysis of SBP.

The measurements will be evaluated while awake in supine position (5 minutes) and subsequently during head up tilt test maneuver (60 degree inclination, 5 minutes). The results of tilt test will be expressed as the change between rest and head up tilt .

Endothelial function Venous endothelial function will be measured by Dorsal Hand Vein technique, previously described by Aellig.

Briefly, a 23-gauge butterfly needle will be inserted into a suitable vein on the back of the hand, with the arm positioned at an upward angle of 30 to allow the complete emptying of veins. A tripod, holding a linear variable differential transformer (LVDT) (Shaevitz Engineering, Pennsuaken, NJ), will be mounted on the back of the hand with the central aperture of the LVDT, containing a movable metal core, at a distance of 10 mm downstream from the dip of the needle. The signal output of the LVDT, which will be linearly proportional to the vertical movement of the core, give a measure of the diameter of the vein. Readings will be taken under a congestive pressure of 40 mm Hg by inflating a blood pressure cuff placed on the upper portion of the arm under study. Results will be presented as normalized dose-response curves in which the diameter of the vein during saline infusion will be defined as 100% dilatation. The vein will be preconstricted to 20% of the baseline size by infusing increasing doses of phenylephrine, a selective A-adrenergic receptor agonist (25-3166 ng/min). The infusion rate of phenylephrine inducing 80% venoconstriction will be kept constant during the entire study, rate, and this degree of constriction will be defined as 0% dilatation for the purpose of subsequent calculations. The vasodilator response expressed in this study will be calculated as a percentage of the range between 0 and 100% dilatation. Drugs will be infused using a Harvard infusion pump (Harvard Apparatus, South Natick, MA) at a flow rate of 0.3 ml/min. After preconstriction of the vein by using phenylephrine, a dose-response curve of acetylcholine (0.36-3600 ng/min) and sodium nitroprusside (50-1000 ng/min) will be constructed with 6 and 2 infusion doses, respectively. Systolic and diastolic BP will be determined before and after each experimental phase with a mercury sphygmomanometer, and heart rate will be measured by the pulse at the radial artery.

Experimental Design The entire study period will be of 12 nights. Using a cross over design the subjects will keep under their usual daily activities and randomized to 5 nights of control sleep or partial sleep deprivation, interposed by 2 nights of wash out (unrestricted sleep). During control period, subjects will be instructed to sleep 8 hours, ranging from a minimal of 7 hours and a maximum of 9 hours and 30 minutes. Partial sleep deprivation will consist of a target sleep between of less than 5 hours, but no less than 3 hours and 30 minutes. Subjects who will not comply with the sleep schedule will be excluded from the final analysis. All measurements described above will be made at the end of control and partial sleep deprivation periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young male volunteers from the urban area of Sao Paulo city

Exclusion Criteria:

* Age less than 21 and more than 45 years
* Body mass index (BMI) >25 kg/m2
* Smoking
* Use of chronic medications and any established medical condition including

  * diabetes mellitus
  * hypertension
  * dyslipidemia
  * heart diseases and
  * sleep disordered breathing

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Venous endothelial function

SECONDARY OUTCOMES:
Sympathetic activity
Inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Josilene L Dettoni, PhD, Principal Investigator — Heart Institute (InCor)
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Dettoni JL, Consolim-Colombo FM, Drager LF, Rubira MC, Souza SB, Irigoyen MC, Mostarda C, Borile S, Krieger EM, Moreno H Jr, Lorenzi-Filho G. Cardiovascular effects of partial sleep deprivation in healthy volunteers. J Appl Physiol (1985). 2012 Jul;113(2):232-6. doi: 10.1152/japplphysiol.01604.2011. Epub 2012 Apr 26. PMID 22539169